CLINICAL TRIAL: NCT04157855
Title: Effectiveness of Abdominal Plane Block (APB) Treatment in the Management and Early Hospital Discharge of Patients Presenting With Acute Exacerbation of Chronic Abdominal Pain (CAP): an Observational Pilot Study
Brief Title: Abdominal Plane Blocks (APB) in Chronic Abdominal Pain (CAP)
Status: Completed | Type: Observational
Sponsor: University Hospitals, Leicester (Other)
Responsible Party: Sponsor
Other Study IDs: 113764
Record Dates: First submitted 2019-11-06; First posted 2019-11-08 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Abdominal Pain; Abdominal Myofascial Pain Syndrome (AMPS); Abdominal Plane Blocks (APB)
MeSH Terms: conditions — Abdominal Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Abdominal Plane Block(s) with depot Steroids — APB Steroids treatment: under real time ultrasound guidance, a 100 mm needle is introduced into the specified plane (subcostal TAP for upper abdomen pain, posterior TAP for lower abdomen pain or TQL for flank and lower abdominal pain). Normal saline (10 ml) is used to open the fascial plane (saline hydrodissection). Then 40 mg of depomedrone diluted in 10 ml of 0.25% levo-bupivacaine is injected into the plane. . A total of 80 mg of depomedrone (steroid) will be used.
  Other Names: Pulsed Radio frequency Treatment to Abdominal Planes

SUMMARY:
Background: Chronic Abdominal Pain (CAP) is the sixth most common cause of hospital admission from any cause in women and the tenth most common cause in men. In the UK, it has been estimated that chronic abdominal pain costs the economy in excess of £100 million per annum. The mechanism of CAP is poorly understood. Patients with acute exacerbation of their CAP have multiple hospital admissions, prolonged length of stay and utilise significant health care resources. These patients have undergone multiple investigations with negative results leading to frustration for both the patient and the clinician. Additional testing and investigations increases costs, patient morbidity and comes with added risks. Patients are discharged once the flare up settles. The investigators have shown that treating patients with steroid injection followed by pulsed radio frequency treatment six months later can reduce the length of stay, repeat hospital admission, improve mood and provide durable pain relief in patients with CAP. The steroid is injected into a specific plane in the abdominal wall and is called abdominal plane block (APB). The investigators currently offer ABP treatment as a standard treatment in the management of patients with CAP.

Aim of the study is to evaluate the effectiveness of Abdominal Plane Block (APB) treatment in reducing hospital readmission over 12 months in patients admitted with exacerbation of CAP

Methods: The proposed study is a prospective, observational pilot study that will be conducted at Leicester General Hospital over 36 months. After providing written consent, adult patients admitted to the hospital with acute exacerbation of CAP will receive two sequential APB treatments (steroid injection followed by pulsed radio frequency treatment) six month apart. If the first treatment with steroid does not provide any benefit, the participants will receive a rescue treatment (trigger point injection with steroids). Participants will be asked to complete questionnaires on pain scores, mood and quality of life. Length of hospital stay, number of hospital re-admission following APB treatment as well as any complication from the APB treatment will be recorded. Participation in the study will end at 12 months following the first APB treatment on completion of relevant questionnaires.

ELIGIBILITY:
Inclusion Criteria:

1. All patients aged over 18 years.
2. Chronic abdominal pain for above 6 months
3. Moderate to severe pain in the abdomen: Baseline NRS >4 (worst pain the last 24 hours)

Exclusion Criteria:

1. Lack of consent, including from those patients who lack mental capacity to give informed consent.
2. Patients with known history of drug allergy to depomedrone
3. Patients with infection at injection site at on day of treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study is based on a cohort of adult patients who are admitted to the hospital with acute exacerbation of chronic abdominal pain.
  Chronic Abdominal Pain is defined as persistent abdominal pain that lasts for more than three months.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2019-01-09 (Actual); Primary Completion 2022-04-08 (Actual); Study Completion 2022-04-08 (Actual)

PRIMARY OUTCOMES:
Primary outcome will be the number of hospital admissions in 12 months following the first Abdominal Plane Block (APB) treatment when compared to 12 months before the first APB treatment | 12 months
  Data will be obtained from an online hospital database (ICE)

CONTACTS AND LOCATIONS:
Overall Officials: Niraj Gopinath, MD, Principal Investigator — University Hospitals, Leicester
Locations (1):
- Leicester General Hospital, Leicester, Leicestershire, United Kingdom

IPD SHARING:
Plan to Share IPD: No